CLINICAL TRIAL: NCT02308969
Title: Neuronal Correlates of Altered States of Consciousness
Acronym: 5HT2A-fMRI
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EKNZ 2014-344
Record Dates: First submitted 2014-11-18; First posted 2014-12-05 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: altered state of consciousness; functional magnetic resonance imaging (fMRI); hallucination; model psychosis; serotonin receptor; LSD
MeSH Terms: conditions — Hallucinations | interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Placebo, LSD (Other): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 1 arm but two treatment conditions in the same subject.
  Interventions: Drug: LSD; Drug: Placebo

INTERVENTIONS:
Drug: LSD — 100ug per os, single dose
  Other Names: Lysergic Acid Diethylamide
Drug: Placebo — Capsules containing mannitol looking identical to LSD

SUMMARY:
The aim of the present study is to assess the neuronal correlates of alterations in waking consciousness pharmacologically induced by a 5-hydroxytryptamine (HT)2A receptor agonist in healthy subjects using functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
Functional neuroimaging may be useful in the diagnosis and characterization of early schizophrenia. However, little is known about how the subjectively experienced alterations in consciousness and perception are related with objective neuroimaging measures. The present study explores the association of subjective alterations and objective imaging findings and will inform us on the neuronal correlates of psychotic states and whether subjective alterations in perception translate into neuronal activation patterns that can be objectively measured in a brain scanner. Therefore, alterations in consciousness will be assessed in 20 healthy subjects using a random order 2-period (normal and altered state of consciousness) cross-over design. Alterations in consciousness will be induced by the hallucinogenic 5-hydroxytryptamine (HT)2A receptor agonist (5-HT2A) receptor agonist lysergic acid diethylamide (LSD).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years
2. Understanding of the German language
3. Understanding the procedures and the risks associated with the study
4. Participants must be willing to adhere to the protocol and sign the consent form
5. Participants must be willing to refrain from taking illicit psychoactive substances during the study.
6. Participants must be willing to drink only alcohol-free liquids and no xanthine-containing liquids (such as coffee, black or green tea, red bull, chocolate) after midnight of the evening before the study session, as well as during the study day.
7. Women of childbearing potential must have a negative pregnancy test at the beginning of the study and before each study session.

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder
3. Psychotic disorder in first-degree relatives
4. Illicit substance use (except tetrahydrocannabinol (THC)-containing products) more than 10 times or any time within the previous month.
5. Pregnant or nursing women.
6. Participation in another clinical trial (currently or within the last 30 days)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
fMRI brain activity | 1 hour
  Associations between fMRI activity (resting state, amygdala-BOLD response to fear and frontoparietal connectivity during working memory processing) and alterations in waking consciousness pharmacologically induced by LSD

SECONDARY OUTCOMES:
Physiological effects (Association of alterations in consciousness and autonomic nervous system reactions (blood pressure, heart rate, pupil size) | 24 hours
  Association of alterations in consciousness and autonomic nervous system reactions (blood pressure, heart rate, pupil size)
Plasma hormone levels (Associations of alterations in consciousness with plasma hormone levels) | 24 hours
  Associations of alterations in consciousness with plasma hormone levels

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, MAS, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland

REFERENCES:
- [Derived] Mueller F, Lenz C, Dolder PC, Harder S, Schmid Y, Lang UE, Liechti ME, Borgwardt S. Acute effects of LSD on amygdala activity during processing of fearful stimuli in healthy subjects. Transl Psychiatry. 2017 Apr 4;7(4):e1084. doi: 10.1038/tp.2017.54. PMID 28375205
- [Derived] Dolder PC, Schmid Y, Steuer AE, Kraemer T, Rentsch KM, Hammann F, Liechti ME. Pharmacokinetics and Pharmacodynamics of Lysergic Acid Diethylamide in Healthy Subjects. Clin Pharmacokinet. 2017 Oct;56(10):1219-1230. doi: 10.1007/s40262-017-0513-9. PMID 28197931
- [Derived] Liechti ME, Dolder PC, Schmid Y. Alterations of consciousness and mystical-type experiences after acute LSD in humans. Psychopharmacology (Berl). 2017 May;234(9-10):1499-1510. doi: 10.1007/s00213-016-4453-0. Epub 2016 Oct 7. PMID 27714429
- [Derived] Dolder PC, Schmid Y, Muller F, Borgwardt S, Liechti ME. LSD Acutely Impairs Fear Recognition and Enhances Emotional Empathy and Sociality. Neuropsychopharmacology. 2016 Oct;41(11):2638-46. doi: 10.1038/npp.2016.82. Epub 2016 Jun 1. PMID 27249781